CLINICAL TRIAL: NCT06194630
Title: Application of 68Ga-labeled ACE2 Targeting Probe PET/CT Imaging in Tracing ACE2 Expression and Diagnosis of Lung Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH ACE2 68Ga-A3
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer; Healthy Human
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-A3 (Experimental): Within 1 week, each participant underwent PET/CT scan after intravenous administration of 68Ga-A3
  Interventions: Drug: 68Ga-A3

INTERVENTIONS:
Drug: 68Ga-A3 — Intravenous injection of 68Ga-A3 with the dosage of 1.5-1.8 MBq (0.04-0.05 mCi)/kg. Tracer doses of 68Ga-A3 will be used to image organs or lesions which expresses ACE2 by PET/CT.

SUMMARY:
In the past three years, as the key protein suggested to be involved in host cell entry of SARS-CoV-2, studies of ACE2 aroused people's attention again. Tracking the expression of ACE2 in vivo is crucial to further understanding of COVID-19, dynamically monitoring the effect of antiviral therapy and the development of related vaccines. It is also expected to further conduct in-depth research on the physiological effects of ACE2 and RAAS, and the mechanism of ACEI/ARB (32). With the development of both molecular imaging agents and related equipment, several ACE2-targeting PET imaging agents have been investigated based on different strategies while some of them were tested in clinical trials. The aim of this study was to intercept key ACE2-binding sites from coronavirus RBD and test their potential as ACE2-targeting PET agents.

ELIGIBILITY:
Inclusion Criteria:

* the ability to provide informed written consent
* a medical history without any ACE2-related comorbidities

Exclusion Criteria:

* liver and renal function dysfunction,
* pregnancy or current lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
standardized uptake value (SUV) | through study completion, an average of 1 year
  comparing the SUVmean of different organs or lesions

SECONDARY OUTCOMES:
Diagnostic performance | through study completion, an average of 1 year
  evaluating the number of lung cancer lesions detected by 68Ga-A3

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Nuclear Medicine, Peking Union Medical College Hopital, Chinese Academy of Medical Science, Beijing
  - Peking Union Medical College Hospital, Beijing